CLINICAL TRIAL: NCT03068845
Title: Arteriovenous Fistula: Conventional Angioplasty vs Drug Eluting Balloon-assisted Maturation Intervention Clinical Trial
Acronym: ACADEMIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACADEMIC_01
Record Dates: First submitted 2017-01-24; First posted 2017-03-03 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Stenosis of Arteriovenous Dialysis Fistula
Keywords: non-maturing arteriovenous fistula; stenosis of arteriovenous fistula; drug-eluting balloon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants, referring physicians, outcomes assessors and data analysis team will be masked. The procedurist will not be masked since it is not possible to perform the procedure without masking. The procedurist will not be involved in outcomes assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug-eluting Balloon Angioplasty (DEBA) (Experimental): After predilatation of the target lesion with conventional balloon angioplasty, a drug-eluting balloon will be inflated to an appropriate inflation pressure, but not exceeding the rated burst pressure of the balloon, for at least a minute.
  Interventions: Device: Drug-eluting balloon angioplasty (DEBA)
- Conventional Balloon Angioplasty (CBA) (Active Comparator): The target lesion will be dilated with a conventional angioplasty balloon to an appropriate inflation pressure, but not exceeding the rated burst pressure of the balloon, for at least a minute.
  Interventions: Device: Conventional Balloon Angioplasty (CBA)

INTERVENTIONS:
Device: Drug-eluting balloon angioplasty (DEBA) — DEBA will be performed after pre-dilatation of the target lesion for subjects allocated to the experimental arm.
  If there is more than 1 stenosis, only the most severe stenosis will be designated the target lesion and treated according to treatment allocation. All other stenoses will be treated with conventional balloon angioplasty.
  High pressure balloon angioplasty may be performed if there is poor angioplasty results (significant residual stenosis of more than 30%).
  All patients will be started on dual antiplatelets (aspirin and clopidogrel) for 1 month after intervention, followed by 5 months of aspirin.
  Other Names: Biotronik Passeo Lux 18
  Arms: Drug-eluting Balloon Angioplasty (DEBA)
Device: Conventional Balloon Angioplasty (CBA) — CBA will be performed for the target lesion for subjects allocated to the active comparator arm.
  If there is more than 1 stenosis, only the most severe stenosis will be designated the target lesion and treated according to treatment allocation. All other stenoses will be treated with conventional balloon angioplasty.
  High pressure balloon angioplasty may be performed if there is poor angioplasty results (significant residual stenosis of more than 30%).
  All patients will be started on dual antiplatelets (aspirin and clopidogrel) for 1 month after intervention, followed by 5 months of aspirin.
  Other Names: Biotronik Passeo
  Arms: Conventional Balloon Angioplasty (CBA)

SUMMARY:
The purpose of this randomised clinical trial is to evaluate the efficacy of drug-eluting balloon compared to conventional balloon in balloon-assisted maturation of non-maturing arteriovenous fistula in adult renal failure patients.

DETAILED DESCRIPTION:
This is a single-centre study, where a total of 124 subjects with non-maturing arteriovenous fistula will be randomised (1:1) to either experimental or active comparator arm. Randomisation will be stratified by location of arteriovenous fistula (above versus below elbow).

Each subject will undergo fistulogram in order to assess eligibility criteria. In the event that there is more than 1 eligible stenosis, the most severe stenosis will be considered the target (study) lesion. All other lesions will be treated in the conventional manner. No coil embolisation of collaterals will be performed in the index treatment.

If the subject is allocated to the experimental arm, the target lesion will be treated with pre-dilatation with a conventional balloon before application of the drug-eluting ballon.

If the subject is allocated to the active comparator arm, the target lesion will be treated with a conventional balloon.

High pressure balloon angioplasty may be performed if there is poor angioplasty results (significant residual stenosis of more than 30%).

All subjects will be prescribed 1 month of dual antiplatelets (aspirin and clopidogrel), followed by 5 months of aspirin.

The duration of the study is 12 months. Follow up visits include:

1. Two-weekly follow up visits in the first 3 months after intervention until the patient is deemed ready for trial cannulation.
2. At 3 months after intervention to assess primary outcome.
3. At 6 months after intervention for a fistulogram
4. At 12 months after intervention for study closure.

ELIGIBILITY:
Inclusion Criteria:

1. Non-maturing upper limb arteriovenous fistula (AVF) created 6-24 weeks ago with any one of the following:

   1. Non-maturing on physical examination, or
   2. Failed initial cannulation, or
   3. Failure to achieve prescribed dialysis within prescribed time frame.
2. Stenosis (>50%) along AVF circuit from anastomosis up to, but not including, the subclavian vein.
3. Successful guidewire crossing of target lesion.
4. >= 21 years old.
5. Informed consent given.
6. Patient willing and able to return for 3 month, 6 month fistulogram and 12 month clinic follow up.

Exclusion Criteria:

1. Thrombosed non-maturing AVF
2. Target lesion is longer than 8 cm
3. Previous endovascular therapy for non-maturation of the trial AVF
4. Baseline systolic blood pressure less than 100 mmHg
5. Non-maturing AVF is not planned to be used for dialysis in the immediate future (e.g. chronic kidney disease not requiring haemodialysis yet)
6. Coagulopathy (prothrombin time or activated partial thromboplastin time >1.5 times the median of normal range) that cannot be managed adequately with periprocedural transfusion
7. Thrombocytopenia (platelet count <50,000 /μL) that cannot be managed adequately with periprocedural transfusion
8. Known allergy to iodinated contrast that cannot be managed adequately with pre-procedure medication
9. Allergy / contraindication to dual anti-platelet therapy (aspirin and clopidogrel or ticlopidine) or paclitaxel
10. Acute infection over proposed puncture site
11. Women who are breastfeeding, pregnant or planning on becoming pregnant during study.
12. Men who are planning on fathering children during the study.
13. Participant with medical conditions which in the opinion of the investigator may cause non-compliance with protocol.
14. Currently participating in an investigational drug, biologic or device trial that may have an impact on the AVF or previous enrollment in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Fistula used successfully for haemodialysis (FUSH) | 3 month
  FUSH is met if the fistula can be used with two-needle cannulation for two-thirds or more of all dialysis runs for 1 month and if it delivers the prescribed dialysis within the prescribed time frame.

SECONDARY OUTCOMES:
Target lesion anatomic success | At the end of index procedure
  Target lesion anatomic success is defined as <30% residual stenosis after angioplasty.
Time from intervention to first successful haemodialysis with two-needle cannulation | Up to 12 months
  Time from intervention to first successful haemodialysis with two-needle cannulation.
Target lesion percent stenosis at 6-month fistulogram | At 6 months
  Percent stenosis of target lesion at 6-month fistulogram
Target lesion restenosis rate at 6-month fistulogram | At 6 months
  The incidence of >50% stenosis of target lesion at 6-month fistulogram
Number of repeat interventions to target lesion at 6 months | At 6 months
  Number of repeat interventions to target lesion at 6 months
Number of repeat interventions to target lesion at 12 months | At 12 months
  Number of repeat interventions to target lesion at 12 months
Number of repeat interventions to access circuit at 6 months | At 6 months
  Number of repeat interventions to access circuit at 6 months
Number of repeat interventions to access circuit at 12 months | At 12 months
  Number of repeat interventions to access circuit at 12 months
Post intervention target lesion patency | Up to 12 months
  Interval from intervention to repeat clinically driven intervention to target lesion
Post intervention access circuit primary patency | Up to 12 months
  Primary patency is defined as the interval from balloon angioplasty until the next access thrombosis or repeated intervention to maintain access function, or until access abandonment if no interval intervention. It ends with treatment of a lesion anywhere within the access circuit, from the arterial inflow to the superior vena cava-right atrial junction.
Post intervention access circuit assisted primary patency | Up to 12 months
  Primary assisted patency is defined as the interval from balloon angioplasty until access thrombosis or a surgical intervention that excludes the treated lesion from the access circuit. Examples include percutaneous treatments of either restenosis/occlusion of the previously treated lesion or a new arterial or venous outflow stenosis/occlusion (excluding access thrombosis). It ends with percutaneous thrombolysis/thrombectomy or simple surgical thrombectomy.
Post-intervention access circuit secondary patency | Up to 12 months
  Secondary patency is defined as the interval after balloon angioplasty until the access is surgically declotted, revised or abandoned because of inability to treat the original lesion, choice of surgeon, transplant, loss to follow-up, etc. Examples include thrombolysis and percutaneous thrombectomy, as well as multiple repetitive treatments.
Complication rates | At 12 months
  Complications will be classified according to the Society of Interventional Radiology Standards of Practice Committee.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Da Zhuang, FRCR, MMed, Principal Investigator — Singapore General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katsanos K, Karnabatidis D, Kitrou P, Spiliopoulos S, Christeas N, Siablis D. Paclitaxel-coated balloon angioplasty vs. plain balloon dilation for the treatment of failing dialysis access: 6-month interim results from a prospective randomized controlled trial. J Endovasc Ther. 2012 Apr;19(2):263-72. doi: 10.1583/11-3690.1. PMID 22545894
- [Background] Lai CC, Fang HC, Tseng CJ, Liu CP, Mar GY. Percutaneous angioplasty using a paclitaxel-coated balloon improves target lesion restenosis on inflow lesions of autogenous radiocephalic fistulas: a pilot study. J Vasc Interv Radiol. 2014 Apr;25(4):535-41. doi: 10.1016/j.jvir.2013.12.014. Epub 2014 Feb 12. PMID 24529550
- [Background] Manninen HI, Kaukanen E, Makinen K, Karhapaa P. Endovascular salvage of nonmaturing autogenous hemodialysis fistulas: comparison with endovascular therapy of failing mature fistulas. J Vasc Interv Radiol. 2008 Jun;19(6):870-6. doi: 10.1016/j.jvir.2008.02.024. Epub 2008 Apr 10. PMID 18503901
- [Background] Shin SW, Do YS, Choo SW, Lieu WC, Choo IW. Salvage of immature arteriovenous fistulas with percutaneous transluminal angioplasty. Cardiovasc Intervent Radiol. 2005 Jul-Aug;28(4):434-8. doi: 10.1007/s00270-003-0211-x. PMID 16001144